CLINICAL TRIAL: NCT05230771
Title: Clinical Outcome of Palliative Surgery After Translational Therapy Versus Maintenance Chemotherapy for Metastatic Gastric Cancer: a Single Center Randomized Controlled Trial
Brief Title: Clinical Outcome of Palliative Surgery After Translational Therapy for Metastatic Gastric Cancer Versus Maintenance Chemotherapy for Metastatic Gastric Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., chief physician, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-24
Record Dates: First submitted 2021-12-05; First posted 2022-02-09 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Gastric Cancer; Surgery; Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palliative surgery after translational therapy (Experimental): After randomization, patients received palliative surgery after translational therapy
  Interventions: Combination Product: Palliative surgery after translational therapy
- Chemotherapy alone (Active Comparator): After randomization, patients received chemotherapy alone
  Interventions: Drug: Chemotheraoy along

INTERVENTIONS:
Combination Product: Palliative surgery after translational therapy — A total, distal, or proximal gastrectomy with D1 lymph node dissection was done depending on tumour after translational therapy .
  location.
  Arms: Palliative surgery after translational therapy
Drug: Chemotheraoy along — Patients receive only the prescribed chemotherapy.
  Arms: Chemotherapy alone

SUMMARY:
This single-center, prospective study was conducted to investigate the efficacy and safety of palliative surgery after translational therapy in the treatment of metastatic gastric cancer. The primary endpoint was 2-year overall survival (OS) rate. Secondary endpoints were median OS, progression-free survival (PFS), 1-year OS, adverse events (AE), severe AE, the quality of life (QOL) and treatment cost.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years
* Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically
* CT/MRI, PET-CT, or laparoscopic exploration should be performed before surgery to confirm the diagnosis of distant metastasis
* Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
* Estimated survival time was over 3 months
* The major organs are functioning normally and meet the following criteria:

  (1) Blood routine examination should meet the requirements (no blood transfusion within 14 days):
  1. HB≥100g/L，
  2. WBC≥3×109/L
  3. ANC≥1.5×109/L，
  4. PLT≥100×109/L； （2）Biochemical tests must meet the following criteria：

  <!-- -->

  1. BIL <1.5×upper limit of normal (ULN)，
  2. ALT and AST<2.5ULN，GPT≤1.5×ULN；
  3. Cr≤1ULN，Ccr >60ml/min
* Fertile women must have taken a pregnancy test (serum) within 7 days prior to enrollment with negative results and be willing to use an appropriate method of contraception during the trial period and 8 weeks after the last trial drug; For men, they should be surgically sterilized or agree to use the appropriate method of contraception during the trial period and 8 weeks after the last administration of the trial drug
* Did not participate in other clinical studies before and during treatment
* Subjects voluntarily joined the study and signed informed consent with good compliance and follow-up

Exclusion Criteria:

* History of other malignant disease within past five years
* History of immunodeficiency, including HIV positive, or other acquired congenital immunodeficiency disease, or a history of organ transplantation and allogeneic bone marrow transplantation
* Accompanied by serious heart, lung, liver and kidney diseases, neuropsychiatric disorders, jaundice or associated severe infection
* Women during pregnancy or breast-feeding
* Subjects had poorly controlled cardiovascular clinical symptoms or diseases, including but not limited to:

  1. NYHA class II or more serious heart failure
  2. unstable angina pectoris
  3. myocardial infarction within 1 year
  4. clinically significant ventricular or ventricular arrhythmias that were poorly controlled without or despite clinical intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival rate | 2 year
  Survival rate of patients in the group from the date of enrollment to 2 years after enrollment